CLINICAL TRIAL: NCT07073521
Title: Developing Evidence-Based Cognitive Approaches to Improve Adjustment to Vision Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Chicago Lighthouse (Other)
Responsible Party: Principal Investigator, Patricia Grant, Ph.D., Chief Research Officer, The Chicago Lighthouse
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WSHF - 2025
Record Dates: First submitted 2025-07-10; First posted 2025-07-18 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Depression, Anxiety; Visual Impairment; Adjustment; Adjustment Disorder With Anxious Mood; Adjustment Disorder With Depressed Mood; Blindness, Acquired; Blindness and Low Vision; Vision Loss
Keywords: Visually impaired; Blind; Vision loss; mental health; CBT; Cognitive-behavioral therapy (CBT); mindfulness; adjustment to vision loss; focus group; pilot test; group therapy
MeSH Terms: conditions — Depression; Anxiety Disorders; Vision Disorders; Blindness; Vision, Low; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot Testing - Assessing Feasibility and Acceptability (Experimental): Participants will be testing an 8-week therapeutic strategy combining cognitive behavioral therapy (CBT) with mindfulness practices tailored for people adjusting to vision loss in a group therapy setting and complete assessments before and after completing the program.
  Interventions: Behavioral: Integrated Cognitive Behavioral Therapy (CBT) & Mindfulness Group Intervention for Adjustment to Vision Loss

INTERVENTIONS:
Behavioral: Integrated Cognitive Behavioral Therapy (CBT) & Mindfulness Group Intervention for Adjustment to Vision Loss — The intervention will be an 8-week integrated group therapy curriculum combining cognitive behavioral therapy (CBT) with mindfulness practices designed for individuals adjusting to vision loss.

SUMMARY:
The goal of this study is to develop and pilot test a therapeutic strategy combining cognitive behavioral therapy (CBT) with mindfulness practices tailored for individuals adjusting to vision loss. The study will begin with focus groups to inform the design of the intervention. Participants will complete brief surveys on their background and experiences with vision loss prior to attending a focus group, and some may be invited to a second session to provide additional feedback before preliminary testing begins. In the pilot phase, participants will attend weekly group therapy sessions using the developed intervention and complete assessments before and after the program, including questions about vision status, demographics, and experiences with vision loss.

DETAILED DESCRIPTION:
The goal of this study is to develop and pilot test an 8-week cognitive behavioral therapy (CBT) & mindfulness curriculum tailored for people adjusting to vision loss. Development of the curriculum during the initial phase of this research will include a thorough review of the literature, input from participant groups, and insights from an expert panel. An initial draft of the curriculum will be developed based on the findings from the literature review. 30-40 Participants will have the opportunity to attend up to two focus group sessions to provide feedback and input on content relevance, feasibility, and acceptability of the curriculum. In the pilot testing phase, 15-20 participants will attend eight weekly group therapy sessions held either in-person or virtually using the developed curriculum and will complete assessments before and after the program. These assessments will include questions about your vision, demographics, and experiences with vision loss, as well as collecting baseline and post-intervention measures prior to undergoing the 8-week pilot testing.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are at least 18 years old
* Experiencing varying degrees of vision loss (e.g. mild, moderate, severe)
* Willingness to participate in the focus group or pilot testing and provide feedback

Exclusion Criteria:

* Individuals with severe cognitive impairment affecting participation
* Congenital blindness
* Recent or current participation in another clinical trial study or medical intervention that may interfere with study results
* Documented or self-reported health condition that may interfere with the outcomes of this study.
* Deemed unfit to participate in the study by the site investigator
* Unwilling and/or unable to participate or provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07-13 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Mean Adaption to Vision Loss (AVL) Scale Score | Assessed at baseline and following the 8-week intervention period
  The AVL is a 24-item self-report questionnaire rated on a 5-point Likert scale. Items assess emotional and psychosocial adjustment to vision loss. Scores range from 1 to 5, with higher scores indicating better adaptation. Some items are reverse-scored.

SECONDARY OUTCOMES:
Change from Baseline in Mean Patient Health Questionnaire (PHQ-9) Score | Assessed at baseline and following the 8-week intervention period
  The Patient Health Questionnaire (PHQ-9) measures average changes in depressive symptoms among participants. PHQ-9 scores range from 0 to 27, with higher scores indicating more severe depression.
Change from Baseline in Mean Generalized Anxiety Disorder (GAD-7) Score | Assessed at baseline and following the 8-week intervention period
  The Generalized Anxiety Disorder 7-item (GAD-7) scale is used to assess the severity of anxiety symptoms. Scores range from 0 to 21, with higher scores indicating more severe anxiety. Each item is scored on a 0-3 Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Research Officer, Principal Investigator — The Chicago Lighthouse
Locations (1):
- The Chicago Lighthouse, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No